CLINICAL TRIAL: NCT06649331
Title: Platform Study of ADC Rechallenge in ADC-treated Metastatic Breast Cancer：A Prospective, Open-label, Multicenter, Phase II Trial
Brief Title: Platform Study of ADC Rechallenge in ADC-treated Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N076
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Advanced Breast Cancer; Metastatic Breast Cancer; Triple Negative Breast Cancer (TNBC); HER2-negative Breast Cancer; Breast Cancer
Keywords: platform trial; adaptive design; antibody-conjugated drugs (ADCs); Bayesian predictive probability
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- A (Experimental): SHR-A1811 (HER2 ADC)
  Interventions: Drug: SHR-A1811
- B (Experimental): SHR-A1921 (TROP2 ADC)
  Interventions: Drug: SHR-A1921
- C (Experimental): SHR-A2009 (HER3 ADC)
  Interventions: Drug: SHR-A2009
- D (Experimental): SHR-A2102 (Nectin4 ADC)
  Interventions: Drug: SHR-A2102
- E (Experimental): SHR-A1811 (HER2 ADC) and Famitinib (VEGFR inhibitor)
  Interventions: Drug: SHR-A1811; Drug: Famitinib
- F (Experimental): SHR-A1811 (HER2 ADC) and Fat Module Formula for Special Medical Purposes (for Medium-Chain Triglyceride Supplementation)
  Interventions: Drug: SHR-A1811; Dietary Supplement: Fat Module Formula for Special Medical Purposes

INTERVENTIONS:
Drug: SHR-A1811 — A HER2-directed ADC, via intravenous (into the vein) infusion per protocol.
  Arms: A; E; F
Drug: SHR-A1921 — A TROP2-directed ADC, via intravenous (into the vein) infusion per protocol.
  Arms: B
Drug: SHR-A2009 — A HER3-directed ADC, via intravenous (into the vein) infusion per protocol.
  Arms: C
Drug: SHR-A2102 — A Nectin4-directed ADC, via intravenous (into the vein) infusion per protocol.
  Arms: D
Drug: Famitinib — A VEGFR inhibitor administered orally per the protocol.
  Arms: E
Dietary Supplement: Fat Module Formula for Special Medical Purposes — This nutritional formulation is composed primarily of medium-chain triglycerides (MCT), which are metabolized by the liver to induce nutritional ketosis, thereby significantly elevating circulating levels of beta-hydroxybutyrate (BHB).
  Arms: F

SUMMARY:
This is a prospective, open-label, multicenter, phase II platform trial. The purpose of this study is to test the safety and effectiveness of the antibody-conjugated drugs (ADCs) in patients with advanced breast cancer who had previously used antibody-conjugated drugs.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicenter, phase II platform trial. The purpose of this study is to test the safety and effectiveness of the antibody-conjugated drugs (ADCs) in patients with advanced breast cancer who had previously received ADCs.

The primary endpoint is objective response rate (ORR). This trial aims to learn whether ADC rechallenge works in treating in ADC-treated metastatic breast cancer and identify which ADC works better for subsets on the basis of molecular characteristics and ADC treatment history of their disease with high ORR. Study drugs involved in this study including but not limited to: SHR-A1811 (HER2 ADC), SHR-A1921 (TROP2 ADC), SHR-A2009 (HER3 ADC) and SHR-A2102 (Nectin 4 ADC).

This platform trial is adaptive design. Novel ADC regimens with sufficiently high activities that show a high Bayesian predictive probability will graduate from the trial with their corresponding biomarker signature(s). ADCs will be dropped if they show a low probability of improved efficacy with any biomarker signature. New ADCs will enter as those that have undergone testing complete their evaluation.

Based on the existing four ADC treatment cohorts on this platform, a maximum of 120 subjects were planned to be enrolled in each ADC treatment cohort. According to the previous ADC treatment history and target, the subjects were randomly assigned to each cohort by adaptive randomization. On the basis of previous clinical data at our center, we limited the enrollment of a minimum of 10 participants per cohort to avoid underrepresentation of any cohort. During the course of the study, ORR will be evaluated periodically for every additional 10 results according to the Bayesian monitoring method, and the proportion of random assignment to each cohort will be adjusted according to the calculated posterior probability using response-adaptive randomization (RAR). Graduation (successful validation) or elimination (failed validation) of ADC rechallenge treatment will be considered according to the posterior probability of an ADC cohort and the data of primary efficacy endpoint, secondary efficacy endpoints and safety endpoints. Additional targeted regimens may be added to the platform regimen as feasible as assessed by the investigators, and the protocol will be modified accordingly at that time.

The efficacy was evaluated by CT or MRI every 6 weeks (±1 week) according to RECIST 1.1. Subjects with CR or PR were required to have radiologic response confirmation at least 4 weeks. Tumor assessments were performed every 9 weeks (±1 week) after 36 weeks of treatment until disease progression, initiation of new antineoplastic therapy, withdrawal of consent, loss to follow-up, death, or the end of the study, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Locally advanced breast cancer (unable to undergo radical local treatment) or recurrent metastatic breast cancer;
3. Previously received ADCs;
4. The most recent pathology results will be considered for enrollment according to local testing of ER, PR and HER2. Participants with any hormone receptor (HR) status will be allowed on study.
5. Prior endocrine therapy: Participants with HR-positive breast cancer must have received prior CDK4/6 inhibitor;
6. Participants must have measurable disease per RECIST 1.1.
7. The functions of the main organs are basically normal and meet the following conditions:

   I. Blood routine examination criteria shall meet: HB ≥90 g/L (no blood transfusion within 14 days); The ANC acuity 1.5 x 10^9 / L; PLT acuity 75 x 10^9 / L; II. Biochemical tests should meet the following criteria: TBIL ≤1.5×ULN (upper limit of normal value); ALT and AST ≤3×ULN; If liver metastases were present, ALT and AST≤ 5×ULN; Serum Cr ≤1.5×ULN, endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula); III. LVEF≥50%
8. They have not received radiotherapy, molecular targeted therapy, or surgery within 3 weeks before the start of the study, and have recovered from the acute toxicity of previous treatment (if surgery was performed, the wound has healed completely); No peripheral neuropathy or grade I peripheral neurotoxicity; Participants may have discontinued all CDK4/6 inhibitor at least 14 days prior to study treatment initiation. Prior endocrine therapy does not require washout.
9. ECOG score ≤2, and life expectancy ≥3 months;
10. Fertile female subjects were required to use a medically approved contraceptive method during the study treatment period and for at least 3 months after the last use of the study drug;
11. Subjects volunteered to join the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Radiotherapy (except for palliative causes), chemotherapy, and immunotherapy were used in the first 3 weeks of treatment, except bisphosphonate (which can be used for bone metastasis);
2. Uncontrolled central nervous system metastases (indicating symptomatic or symptomatic treatment with glucocorticoids or mannitol);
3. A history of clinically important or uncontrolled heart disease, including congestive heart failure, angina pectoris, myocardial infarction, or ventricular arrhythmia within the last 6 months;
4. Presence of the third space effusion (such as massive ascites, pleural effusion, pericardial effusion) that cannot be controlled by drainage or other methods;
5. Participants with who had used immunosuppressive agents or systemic corticosteroids within 2 weeks before the first dose (dose> 10mg/day prednisone or other corticosteroids at the physiological dose of the drug), excluding nasal spray or inhaled corticosteroids;
6. Presence of any active autoimmune disease or a history of autoimmune disease with potential relapse;
7. Known human immunodeficiency virus (HIV) infection that is not well controlled;
8. Known active hepatitis B (HBV DNA≥2000 IU/mL or 104 copies/mL) and hepatitis C (positive for hepatitis C antibodies and HCV-RNA above the lower detection limit of the assay);
9. Persistent grade 1 or higher adverse reactions caused by previous treatments. The exception to this is hair loss or something the researchers don't think should be ruled out. Such cases should be clearly documented in the investigator's notes;
10. Underwent major surgery (except minor outpatient procedures, such as placement of vascular access) within 3 weeks of the first course of trial treatment;
11. Pregnant or lactating patients;
12. Malignancy (except basal cell carcinoma of the skin, which has been cured, and carcinoma in situ of the cervix) in the past 5 years;
13. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study agent or accompanying supportive medications;
14. Serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participating in the study or interfere with the study results
15. Deemed by the investigator to be ineligible for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | The observation period related to this endpoint is up to 36 months.
  Objective response rate (ORR), defined as best overall response of either complete or partial response, will be assessed among participants who start protocol therapy and have measurable disease at screening. Radiographic response will be assessed using RECIST 1.1 criteria as defined per protocol.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | The observation period related to this endpoint is up to 36 months.
  PFS based on Kaplan-Meier methodology will be defined as the time from randomization until the identification of disease progression or death, whichever occurs first. Subjects without disease progression or death at the time of analysis will be censored at the date of last disease evaluation.
Clinical Benefit Rate (CBR) | The observation period related to this endpoint is up to 36 months.
  Clinical Benefit Rate (CBR) is defined as the proportion of participants with CR, PR and stable disease (SD) for ≥ 24 weeks as the best overall response.
Duration of Response (DOR) | The observation period related to this endpoint is up to 36 months.
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause). Participants without reported events are censored at the last disease evaluation.
Overall Survival (OS) | The observation period related to this endpoint is up to 5 years.
  Overall survival based on the Kaplan-Meier method is defined as the time from randomization to death. Participants alive are censored at the last date of contact (including lost-to-follow-up) or at the date of withdrawal of consent, if relevant.
Treatment-Related Toxicity Rate | The observation period related to this endpoint is up to 36 months.
  The percentage of participants who experienced any grade treatment-related adverse event based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms.

OTHER OUTCOMES:
Exploration of translational research markers | The observation period related to this endpoint is up to 36 months.
  The collected subjects' tumor tissues, paracancerous tissues, blood, and fecal samples will be used for discovering exploratory biomarkers (including but not limited to the expression of HER2, TROP2, HER3, Nectin4, etc.). The relationships between discovered biomarkers and subjects' disease status and treatment responses will also be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, M.D., Principal Investigator — Fudan University
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No